CLINICAL TRIAL: NCT00239811
Title: A Two-year Extension to a One-year, Multicenter, Partially Blinded, Double Dummy, Randomized Study to Evaluate the Efficacy and Safety of FTY720 Combined With Reduced-dose or Full-dose Cyclosporine, USP [Modified] (Novartis Brand) and Corticosteroids Versus Mycophenolate Mofetil Combined With Full-dose Cyclosporine, USP [Modified] (Novartis Brand) and Corticosteroids, in de Novo Adult Renal Transplant Recipients
Brief Title: Long Term Efficacy and Safety of FTY720 in de Novo Adult Renal Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720A0124E1
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Renal Transplantation
Keywords: Transplantation, kidney, and organ transplant.
MeSH Terms: interventions — Fingolimod Hydrochloride

INTERVENTIONS:
Drug: FTY720

SUMMARY:
This study will evaluate the long term safety and efficacy of FTY720 combined with cyclosporine and corticosteroids in patients receiving a kidney organ transplant

ELIGIBILITY:
Inclusion Criteria

* Patients who completed the 12 month core study
* Patients who gave written informed consent to participate in the study Exclusion Criteria
* Not applicable Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 684
Dates: Start 2004-04; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
IA, IB, IIA, IIB, III, or humoral rejection diagnosed by biopsy according to Banff 97 criteria within 36 months post transplant
Permanent resumption of dialysis within 36 months post transplant
Surgical removal of graft within 36 months post transplant
Death within 36 months post transplant
Withdrawal of consent, death, or lost to follow up within 36 months post transplant
Serum creatinine, calculated creatinine clearance and urine-protein/creatinine ratio at Months 18, 24, 30 and 36
FEV1 , FVC, FEV1/FVC, DLCO and FEF 25%-75% at Months 18, 24, 30 and 36
Absolute lymphocyte count at Months 18, 24, 30 and 36.

SECONDARY OUTCOMES:
Physical examinations at Months 18, 24, 30 and 36
Vital signs at Months 18, 24, 30 and 36
Electrocardiogram at Months 24 and 36
Chest X-ray Months 24 and 36
Safety laboratory tests 18, 24, 30 and 36
Ophthalmic evaluations 18, 24, 30 and 36
AEs and SAEs
FTY720/CsA levels at Months 18, 24, 30 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis